CLINICAL TRIAL: NCT04114799
Title: A Comparison of Perioperative Fluid Management Using Invasive Haemodynamical Measurement of Fluid Responsiveness (Aisys GE) and Non-invasive Measurement of Haemodynamics (ClearSight System, Edwards) During Brain Surgery
Brief Title: Haemodynamical Optimization During Brain Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, principal investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHradec Kralove
Record Dates: First submitted 2019-09-07; First posted 2019-10-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Brain Edema
Keywords: fluid responsiveness; haemodynamical monitoring; ClearSight
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A invasive haemodynamical measurement (Active Comparator): No continuous infusion of fluids will be used intraoperatively. A defined amount of fluid (20 ml of Plasmalyte, Baxter) will be used to flush the anesthetics and other drugs only. Fluid bolus will be applied in case of protocol defined hypotension according to the value of systolic pressure variation SPV (Aisys GE). The value of SPV (tidal volume 6 ml/kg) above 8% will be used to predict fluid responsiveness. In case of fluid responsiveness, bolus of 2ml/kg of Plasmalyte will be given within 10 minutes. Boluses will be repeated in hypotensive patients if fluid responsiveness persists. Norepinephrine will be used in hypotensive patients without predicted fluid responsiveness.
  Interventions: Procedure: Hemodynamic management based on invasive fluid responsiveness parameters
- Group B non-invasive haemodynamical measurement (Experimental): No continuous infusion of fluids will be used intraoperatively. A defined amount of fluid (20 ml of Plasmalyte, Baxter) will be used to flush the anesthetics and other drugs only. Fluid management and the use of norepinephrine will follow a protocol based on the values of cardiac index level, systemic vascular resistance and systolic volume variation (SVV) (ClearSight, Edwards).
  Interventions: Procedure: Hemodynamic management based on noninvasive cardiac output and SVV measurement

INTERVENTIONS:
Procedure: Hemodynamic management based on invasive fluid responsiveness parameters — In case of hypotension (reduction of MAP for more than 15% of individual blood pressure) the SPV value more than 8% will be used as a trigger for the bolus of 2 ml/kg of Plasmalyte (Baxter)
  Arms: Group A invasive haemodynamical measurement
Procedure: Hemodynamic management based on noninvasive cardiac output and SVV measurement — In case of hypotension (reduction of MAP for more than 15% of individual blood pressure) the systemic vascular resistance (SVR) value will be used to trigger norepinephrine infusion. In patients with low SVR norepinephrine infusion will be started. In patients with high SVR value either fluid bolus (in patient with SVV value above 8%), or dobutamine infusion (in patients with SVV value below or equal 8%) will be used.
  Arms: Group B non-invasive haemodynamical measurement

SUMMARY:
The decision to give fluids perioperatively could be based on methods used to identify preload responsiveness, either invasive or noninvasive estimates of stroke volume variation during mechanical ventilation. This study compares fluid management using invasive measurement SPV/PPV (Aisys GE) and noninvasive haemodynamic measurement (ClarSight, Edwards).

DETAILED DESCRIPTION:
The aim of the study is to optimise fluid management and to reduce perioperative risks during brain surgery. Adequate perioperative management guided by hemodynamic monitoring can help to reduce the risk of complications and thus potentially improve outcomes.

This study compares fluid management algorithms based either on invasive detection of fluid responsiveness using pulse pressure variation (PPV) and systolic pressure variation (SPV) values (Aisys GE monitoring system) in group A, or on noninvasive measurement of haemodynamics (stroke volume variation (SVV), cardiac index (CI) and systemic vascular resistance (SVR) values) (ClearSight, Edwards) in group B.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma scale 15
* ASA Physical Status Classification System I-III
* planed surgery for brain tumor to 5 hours
* postoperative awakening
* sinus rhythm

Exclusion Criteria:

* NYHA III, IV
* BMI over 40 in females and over 35 in men
* awake operation
* postoperative artificial ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
fluid balance difference | up to 5 hours after start of operation
  the difference between fluid intake and output and losses during surgery will be calculated

SECONDARY OUTCOMES:
mean dose of norepinephrine | up to 5 hours after start of operation
  mean dose of norepinephrine will be calculated from total delivered dose devided by time of the surgery
level of creatinin | 24 hours
  plasma level of creatinin measured on the first postoperative day
postoperative lung dysfunction | 1 day
  postoperative lung dysfunction defined as SpO2 value less than 92% or oxygen therapy more than 6 hours postoperatively
length of postoperative stay | up to 2 month after surgery
  number of days of stay in the hospital after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Dostal, MD, Ph.D., Study Director — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia